CLINICAL TRIAL: NCT06112743
Title: MEMENTO - A Phase 4, Single-arm, Open-label Clinical Study to Evaluate Mavacamten in Adults With Symptomatic Obstructive Hypertrophic Cardiomyopathy to Assess the Impact on Myocardial Structure With Cardiac Magnetic Resonance Imaging (CMR)
Brief Title: A Study to Evaluate Mavacamten Impact on Myocardial Structure in Participants With Symptomatic Obstructive Hypertrophic Cardiomyopathy
Acronym: MEMENTO
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV027-1088
Record Dates: First submitted 2023-10-27; First posted 2023-11-01 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cardiomyopathy, Hypertrophic
Keywords: BMS-986427; MYK-461; Mavacamten; Obstructive Hypertrophic Cardiomyopathy (oHCM); Camyzos; Cardiac Magnetic Resonance Imaging (CMR)
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mavacamten (Experimental)
  Interventions: Drug: Mavacamten

INTERVENTIONS:
Drug: Mavacamten — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the mavacamten impact on myocardial structure with cardiac magnetic resonance imaging (CMR) in adult participants with symptomatic obstructive hypertrophic cardiomyopathy (oHCM) [New York Heart Association (NYHA) Functional Class II or III].

ELIGIBILITY:
Inclusion Criteria

* Diagnosed with obstructive hypertrophic cardiomyopathy (oHCM), in accordance with current American College of Cardiology Foundation/American Heart Association and European Society of Cardiology guidelines as below:.
* Left ventricular outflow tract (LVOT) peak gradient ≥ 30 mmHg and ≥ 50 mmHg after Valsalva or after exercise.
* Left ventricular ejection fraction (LVEF) ≥ 55% at rest.
* New York Heart Association (NYHA) functional class II or III symptoms.

Exclusion Criteria

* A known infiltrative or storage disorder causing cardiac hypertrophy that mimics oHCM.
* Documented obstructive coronary artery disease or history of myocardial infarction.
* A history of resuscitated sudden cardiac arrest or life-threatening ventricular arrhythmia within 6 months prior to screening.
* An implantable cardioverter defibrillator (ICD) or pacemaker, or another contraindication for cardiac magnetic resonance imaging (CMR).
* Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2026-07-09 (Estimated); Study Completion 2026-07-09 (Estimated)

PRIMARY OUTCOMES:
Composite of maximum left atrial volume index (LAVI) and left ventricular mass index (LVMI) at Week 48 | At week 48
  Participants achieving both of the following criteria at Week 48 cardiac magnetic resonance imaging (CMR) assessment:
  * A decrease of at least 5 mL/m2 in maximum LAVI from baseline
  * A decrease of at least 5 g/m2 in LVMI from baseline

SECONDARY OUTCOMES:
Proportion of participants who had at least 1 class of improvement from baseline in New York Heart Association (NYHA) class at Week 48 | At week 48
Change from baseline in maximum left atrial volume index (LAVI) at Week 48 | At week 48
Change from baseline in left ventricular mass index (LVMI) at Week 48 | At week 48
Incidence of major adverse cardiac events (MACE) | Up to 48 weeks
Incidence of MACE-expanded events | Up to 48 weeks
All-cause mortality | Up to 48 weeks
Incidence of heart failure (HF) events | Up to 48 weeks
Incidence of HF events with systolic dysfunction | Up to 48 weeks
Incidence of atrial fibrillation (AF)/atrial flutter | Up to 48 weeks
Incidence of cardiovascular (CV) mortality | Up to 48 weeks
Incidence of ventricular tachyarrhythmias | Up to 48 weeks
Incidence of nonvasovagal syncope and seizures | Up to 48 weeks
Incidence of treatment emergent adverse events (TEAEs) | Up to 48 weeks
Severity of TEAEs | Up to 48 weeks
Incidence of treatment emergent serious adverse events (SAEs) | Up to 48 weeks
TEAEs leading to discontinuation from study intervention | Up to 48 weeks
TEAEs leading to laboratory abnormalities | Up to 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (23):
- United States (7):
  - Local Institution - 0087, West Hollywood, California
  - Local Institution - 0003, Atlanta, Georgia
  - Local Institution - 0093, Boston, Massachusetts
  - Local Institution - 0090, Cleveland, Ohio
  - Local Institution - 0086, Pittsburgh, Pennsylvania
  - Local Institution - 0017, Houston, Texas
  - Local Institution - 0035, Murray, Utah
- Argentina (6):
  - Local Institution - 0076, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0075, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0079, Pilar, Buenos Aires
  - Local Institution - 0077, Córdoba, Córdoba Province
  - Local Institution - 0074, Rosario, Santa Fe Province
  - Local Institution - 0080, Buenos Aires
- Australia (3):
  - Local Institution - 0015, Camperdown, New South Wales
  - Local Institution - 0085, Chermside, Queensland
  - Local Institution - 0005, Melbourne, Victoria
- Canada (2):
  - Local Institution - 0001, Montreal, Quebec
  - Local Institution - 0068, Québec, Quebec
- Switzerland (4):
  - Local Institution - 0058, Lucerne, Luzern (de)
  - Local Institution - 0029, Lugano, Ticino (it)
  - Local Institution - 0061, Geneva
  - Local Institution - 0024, Zürich (de)
- Local Institution - 0025, Leeds, Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06112743.html